CLINICAL TRIAL: NCT01120704
Title: Project 3: Identifying Optimal Strategies of Increasing Smokers' Adherence to Cessation Medications
Brief Title: Evaluation of Treatments to Improve Smoking Cessation Medication Adherence
Acronym: Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Dean Health System (Other); Mercy Health System (Network); Wake Forest University Health Sciences (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H-2010-0049; 9P50CA143188 (NIH)
Record Dates: First submitted 2010-05-03; First posted 2010-05-11 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Smoking; Smoking Cessation; Adherence; Nicotine Dependence; Motivation
Keywords: Smoking; Smoking Cessation; Adherence; Nicotine; Motivation
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder | interventions — Transdermal Patch; Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (32):
- 1, 26Wks, Counseling, CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Automated Adherence Prompting Phone Calls
- 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 4, 26Wks, Counseling, CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM)
- 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 6, 26Wks, Counseling, No CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Automated Adherence Prompting Phone Calls
- 7, 26Wks, Counseling, No CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 8, 26Wks, Counseling, No CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling
- 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 10, 26Wks, No Counseling, CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Automated Adherence Prompting Phone Calls
- 11, 26Wks, No Counseling, CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 12, 26Wks, No Counseling, CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM)
- 13, 26Wks, No Counseling, No CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 14, 26Wks, No Counseling, No CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Automated Adherence Prompting Phone Calls
- 15, 26Wks, No Counseling, No CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 16, 26Wks, No Counseling, No CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  26Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum)
- 17, 8Wks, Counseling, CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Automated Adherence Prompting Phone Calls
- 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 20, 8Wks, Counseling, CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Cognitive Medication Adherence Counseling (CAM)
- 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 22, 8Wks, Counseling, No CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Automated Adherence Prompting Phone Calls
- 23, 8Wks, Counseling, No CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling; Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 24, 8Wks, Counseling, No CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Intensive Maintenance Counseling
- 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 26, 8Wks, No Counseling, CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Automated Adherence Prompting Phone Calls
- 27, 8Wks, No Counseling, CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 28, 8Wks, No Counseling, CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Cognitive Medication Adherence Counseling (CAM)
- 29, 8Wks, No Counseling, No CAM, AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback; Behavioral: Automated Adherence Prompting Phone Calls
- 30, 8Wks, No Counseling, No CAM, AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Automated Adherence Prompting Phone Calls
- 31, 8Wks, No Counseling, No CAM, No AutoCalls, Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device + Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum); Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback
- 32, 8Wks, No Counseling, No CAM, No AutoCalls, No Feedback (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?:
  8Wks Medication duration during quit attempt, No Maintenance Counseling, No Cognitive Adherence Intervention, No Automated Medication Adherence Calls, Electronic Medication Monitoring Device but No Feedback
  Interventions: Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum)

INTERVENTIONS:
Drug: Short Term Combination Nicotine Replacement Therapy (patch + gum) — IF participant smokes >10 cigs/day AND is randomized to a 8 week condition: they will be asked to take one 21 mg patch/day for 4 weeks, THEN one 14 mg patch/day for 2 weeks, THEN one patch 7mg/day for 2 weeks.Participants will also be asked to use 4-mg gum every 1-2 hours (9 pieces maximum per day)for 6 weeks and decrease gum use over the 2 weeks prior to medication termination until down to one gum piece every 4-8 hours by the last week of treatment.
  IF participant smokes 5-10 cigs/day AND is randomized to the 8 week medication condition: they will be asked to take one 14 mg patch/day for 4 weeks, THEN one 7 mg patch/day for 4 weeks. Participants will also be asked to use 2-mg gum every 1-2 hours (9 pieces max per day)for 6 weeks and decrease gum use over the 2 weeks prior to medication termination until down to one gum piece every 4-8 hours by the last week of treatment.
  Arms: 17, 8Wks, Counseling, CAM, AutoCalls, Feedback; 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback; 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback; 20, 8Wks, Counseling, CAM, No AutoCalls, No Feedback; 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback; 22, 8Wks, Counseling, No CAM, AutoCalls, No Feedback; 23, 8Wks, Counseling, No CAM, No AutoCalls, Feedback; 24, 8Wks, Counseling, No CAM, No AutoCalls, No Feedback; 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback; 26, 8Wks, No Counseling, CAM, AutoCalls, No Feedback; 27, 8Wks, No Counseling, CAM, No AutoCalls, Feedback; 28, 8Wks, No Counseling, CAM, No AutoCalls, No Feedback; 29, 8Wks, No Counseling, No CAM, AutoCalls, Feedback; 30, 8Wks, No Counseling, No CAM, AutoCalls, No Feedback; 31, 8Wks, No Counseling, No CAM, No AutoCalls, Feedback; 32, 8Wks, No Counseling, No CAM, No AutoCalls, No Feedback
Drug: Long Term Combination Nicotine Replacement Therapy (patch + gum) — IF the participant smokes >10 cigs/day AND is randomized to a 26 week medication condition: they will be asked to take one 21 mg patch per day for 22 weeks, THEN one 14 mg patch per day for 2 weeks, THEN one patch 7 mg patch per day for 2 weeks. Participants will also be asked to use one piece of one 4-mg- gum every 1-2 hours (9 pieces maximum per day)for 24 weeks and decrease gum use over the 2 weeks prior to medication termination until they are down to one gum piece every 4-8 hours by the last week of treatment.
  IF the participant smokes 5-10 cigs/day AND is randomized to a 26 week medication condition: they will be asked to take one 14 mg patch per day for 22 weeks, THEN one patch 7 mg patch per day for 4 weeks. Participants will also be asked to use one piece of 2-mg gum every 1-2 hours (9 pieces maximum per day)for 24 weeks and decrease gum use over the 2 weeks prior to medication termination until they are down to one gum piece every 4-8 hours by the last week of treatment.
  Arms: 1, 26Wks, Counseling, CAM, AutoCalls, Feedback; 10, 26Wks, No Counseling, CAM, AutoCalls, No Feedback; 11, 26Wks, No Counseling, CAM, No AutoCalls, Feedback; 12, 26Wks, No Counseling, CAM, No AutoCalls, No Feedback; 13, 26Wks, No Counseling, No CAM, AutoCalls, Feedback; 14, 26Wks, No Counseling, No CAM, AutoCalls, No Feedback; 15, 26Wks, No Counseling, No CAM, No AutoCalls, Feedback; 16, 26Wks, No Counseling, No CAM, No AutoCalls, No Feedback; 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback; 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback; 4, 26Wks, Counseling, CAM, No AutoCalls, No Feedback; 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback; 6, 26Wks, Counseling, No CAM, AutoCalls, No Feedback; 7, 26Wks, Counseling, No CAM, No AutoCalls, Feedback; 8, 26Wks, Counseling, No CAM, No AutoCalls, No Feedback; 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback
Behavioral: Intensive Maintenance Counseling — Participants randomized to this condition will receive eight 15-minute phone counseling sessions at Weeks 3, 4, 6, 8, 10, 14, 18 & 22. The counseling will encourage continued practice of coping skills, and avoidance of danger situations. Another emphasis will be the continued provision of social support as a means of enhancing motivation. Participants who have relapsed will receive counseling aimed at motivating and planning renewed quit attempts. Other aims are enhancing motivation, especially competence self-appraisals, providing intratreatment support, and encouraging pleasurable activities.
  Arms: 1, 26Wks, Counseling, CAM, AutoCalls, Feedback; 17, 8Wks, Counseling, CAM, AutoCalls, Feedback; 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback; 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback; 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback; 20, 8Wks, Counseling, CAM, No AutoCalls, No Feedback; 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback; 22, 8Wks, Counseling, No CAM, AutoCalls, No Feedback; 23, 8Wks, Counseling, No CAM, No AutoCalls, Feedback; 24, 8Wks, Counseling, No CAM, No AutoCalls, No Feedback; 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback; 4, 26Wks, Counseling, CAM, No AutoCalls, No Feedback; 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback; 6, 26Wks, Counseling, No CAM, AutoCalls, No Feedback; 7, 26Wks, Counseling, No CAM, No AutoCalls, Feedback; 8, 26Wks, Counseling, No CAM, No AutoCalls, No Feedback
Behavioral: Cognitive Medication Adherence Counseling (CAM) — Participants randomized to this condition will be given a brief (10 minute) session of CAM treatment at both Visits 1 and 2. CAM will include information on NRT such as the following: NRT reduces withdrawal and urges; sustained use reduces the likelihood of relapse; willpower and medication make a good combination; NRT will help a lapsing smoker reachieve abstinence. The tailored counseling component of the CAM intervention is based on brief evaluation of the smoker's beliefs, concerns, and possible misconceptions about smoking cessation medications.
  Arms: 1, 26Wks, Counseling, CAM, AutoCalls, Feedback; 10, 26Wks, No Counseling, CAM, AutoCalls, No Feedback; 11, 26Wks, No Counseling, CAM, No AutoCalls, Feedback; 12, 26Wks, No Counseling, CAM, No AutoCalls, No Feedback; 17, 8Wks, Counseling, CAM, AutoCalls, Feedback; 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback; 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback; 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback; 20, 8Wks, Counseling, CAM, No AutoCalls, No Feedback; 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback; 26, 8Wks, No Counseling, CAM, AutoCalls, No Feedback; 27, 8Wks, No Counseling, CAM, No AutoCalls, Feedback; 28, 8Wks, No Counseling, CAM, No AutoCalls, No Feedback; 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback; 4, 26Wks, Counseling, CAM, No AutoCalls, No Feedback; 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback
Behavioral: Electronic Medication Monitoring Device (the Helping Hand) + Feedback — If randomized to this condition, the case manager will give patients a computer-generated feedback sheet showing the patient's medication self-administration since the last visit. The case manager will provide problem-solving counseling regarding barriers to medication use. This problem-solving counseling intervention will be given in brief in-person sessions (three in-person sessions for those in the 8 week medication condition and five in-person sessions for those in the 26 week medication condition). Medication monitoring counseling will also occur via phone (two 10-minute sessions for those in the 8 week medication condition and four 10-minute sessions for those in the 26 week medication condition).
  Arms: 1, 26Wks, Counseling, CAM, AutoCalls, Feedback; 11, 26Wks, No Counseling, CAM, No AutoCalls, Feedback; 13, 26Wks, No Counseling, No CAM, AutoCalls, Feedback; 15, 26Wks, No Counseling, No CAM, No AutoCalls, Feedback; 17, 8Wks, Counseling, CAM, AutoCalls, Feedback; 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback; 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback; 23, 8Wks, Counseling, No CAM, No AutoCalls, Feedback; 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback; 27, 8Wks, No Counseling, CAM, No AutoCalls, Feedback; 29, 8Wks, No Counseling, No CAM, AutoCalls, Feedback; 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback; 31, 8Wks, No Counseling, No CAM, No AutoCalls, Feedback; 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback; 7, 26Wks, Counseling, No CAM, No AutoCalls, Feedback; 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback
Behavioral: Automated Adherence Prompting Phone Calls — Participants in this condition will receive fully automated prompts with messages designed to encourage participants to take their medication.
  Adherence prompting calls will occur two times in the first week of the quit attempt, and then once a week in weeks 2, 3, 4, 5, and 7. Those in the 26-Week medication condition who are assigned to the active adherence prompting calls intervention, will receive one prompting call a week during Weeks 11, 15, 19 & 23.
  Arms: 1, 26Wks, Counseling, CAM, AutoCalls, Feedback; 10, 26Wks, No Counseling, CAM, AutoCalls, No Feedback; 13, 26Wks, No Counseling, No CAM, AutoCalls, Feedback; 14, 26Wks, No Counseling, No CAM, AutoCalls, No Feedback; 17, 8Wks, Counseling, CAM, AutoCalls, Feedback; 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback; 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback; 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback; 22, 8Wks, Counseling, No CAM, AutoCalls, No Feedback; 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback; 26, 8Wks, No Counseling, CAM, AutoCalls, No Feedback; 29, 8Wks, No Counseling, No CAM, AutoCalls, Feedback; 30, 8Wks, No Counseling, No CAM, AutoCalls, No Feedback; 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback; 6, 26Wks, Counseling, No CAM, AutoCalls, No Feedback; 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback

SUMMARY:
Many smokers fail to take their smoking cessation medication as recommended. This research is designed to identify treatments that improve the use of cessation medications and to determine whether an increase in medication use results in increased cessation success. This research will also identify treatments that help people stay quit after a quit attempt and will pioneer more efficient research methods.

DETAILED DESCRIPTION:
Nonadherent use of smoking cessation medications is very common and highly associated with cessation failure. However, little is presently known about how to improve adherence and whether improved adherence will actually boost cessation success (i.e., its causal role is unknown). This research represents groundbreaking integration of 1) basic theory and data on tobacco dependence, adherence, and intervention mechanisms with 2) the state-of-the-art Intervention Optimization Cycle methodology. This methodology uses factorial designs to efficiently engineer and evaluate intervention components, and to develop an optimal comprehensive treatment package. Participants in Project 3 will be smokers (N = 544) visiting primary care clinics for a regular outpatient visit who, when asked, express an interest in quitting and agree to participate in a smoking cessation research study. The experiment will comprise five experimental factors (2X2X2X2X2), and participants will have a 50% chance of being assigned one of the levels of each factor. The five factors include one medication factor (medication duration: 8 vs. 26 weeks), one counseling factor (maintenance counseling vs. no maintenance counseling), and three adherence factors: 1) Cognitive Medication Adherence Counseling (C-MAC); C-MAC vs. no C-MAC; 2) electronic medication monitoring device (the Helping Hand) + Feedback vs. the medication monitoring device alone; and 3) automated adherence prompting phone calls vs. no prompting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Report smoking at least 5 cigarettes per day for the previous 6 months;
* Able to read and write English;
* Agree to attend visits, to respond to coaching calls, and to respond to Interactive Voice Response (IVR) phone prompts;
* Plans to remain in the intervention catchment area for at least 12 months;
* Currently interested in quitting smoking (defined as would like to try to quit in the next 30 days).
* All women of childbearing potential will be required to agree to use an acceptable method of birth control to prevent pregnancy during the study.

Exclusion Criteria:

* Currently taking bupropion, Wellbutrin, chantix or varenicline (current use of NRT is not exclusionary if the participant agrees to use only study medication for the duration of the study);
* Study candidate is pregnant, trying to get pregnant, or nursing.
* A history of psychosis or bipolar disorder
* A history of skin or allergic reactions while using a nicotine patch.
* Had a heart attack, stroke, or abnormal electrocardiogram within the past 4 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD, MPH, MBA, Principal Investigator — University of Wisconsin School of Medicine and Public Health, Center for Tobacco Research and Intervention; Tanya R Schlam, PhD, Study Director — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Background] McCarthy DE, Piasecki TM, Lawrence DL, Jorenby DE, Shiffman S, Baker TB. Psychological mediators of bupropion sustained-release treatment for smoking cessation. Addiction. 2008 Sep;103(9):1521-33. doi: 10.1111/j.1360-0443.2008.02275.x. PMID 18783504
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Schlam TR, Baker TB, Smith SS, Bolt DM, McCarthy DE, Cook JW, Hayes-Birchler T, Fiore MC, Piper ME. Electronically Monitored Nicotine Gum Use Before and After Smoking Lapses: Relationship With Lapse and Relapse. Nicotine Tob Res. 2020 Oct 29;22(11):2051-2058. doi: 10.1093/ntr/ntaa116. PMID 32598468
- [Derived] Schlam TR, Cook JW, Baker TB, Hayes-Birchler T, Bolt DM, Smith SS, Fiore MC, Piper ME. Can we increase smokers' adherence to nicotine replacement therapy and does this help them quit? Psychopharmacology (Berl). 2018 Jul;235(7):2065-2075. doi: 10.1007/s00213-018-4903-y. Epub 2018 Apr 25. PMID 29696311
- See also: University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1, 26Wks, Counseling, CAM, AutoCalls, Feedback | 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback | 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback | 4, 26Wks, Counseling, CAM, No AutoCalls, No Feedback | 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback | 6, 26Wks, Counseling, No CAM, AutoCalls, No Feedback | 7, 26Wks, Counseling, No CAM, No AutoCalls, Feedback | 8, 26Wks, Counseling, No CAM, No AutoCalls, No Feedback | 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback | 10, 26Wks, No Counseling, CAM, AutoCalls, No Feedback | 11, 26Wks, No Counseling, CAM, No AutoCalls, Feedback | 12, 26Wks, No Counseling, CAM, No AutoCalls, No Feedback | 13, 26Wks, No Counseling, No CAM, AutoCalls, Feedback | 14, 26Wks, No Counseling, No CAM, AutoCalls, No Feedback | 15, 26Wks, No Counseling, No CAM, No AutoCalls, Feedback | 16, 26Wks, No Counseling, No CAM, No AutoCalls, No Feedback | 17, 8Wks, Counseling, CAM, AutoCalls, Feedback | 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback | 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback | 20, 8Wks, Counseling, CAM, No AutoCalls, No Feedback | 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback | 22, 8Wks, Counseling, No CAM, AutoCalls, No Feedback | 23, 8Wks, Counseling, No CAM, No AutoCalls, Feedback | 24, 8Wks, Counseling, No CAM, No AutoCalls, No Feedback | 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback | 26, 8Wks, No Counseling, CAM, AutoCalls, No Feedback | 27, 8Wks, No Counseling, CAM, No AutoCalls, Feedback | 28, 8Wks, No Counseling, CAM, No AutoCalls, No Feedback | 29, 8Wks, No Counseling, No CAM, AutoCalls, Feedback | 30, 8Wks, No Counseling, No CAM, AutoCalls, No Feedback | 31, 8Wks, No Counseling, No CAM, No AutoCalls, Feedback | 32, 8Wks, No Counseling, No CAM, No AutoCalls, No Feedback
Started | 13 | 17 | 14 | 19 | 16 | 19 | 15 | 15 | 22 | 20 | 17 | 16 | 17 | 19 | 18 | 18 | 14 | 16 | 17 | 18 | 17 | 16 | 21 | 16 | 18 | 14 | 18 | 18 | 19 | 15 | 14 | 18
Completed | 10 | 13 | 13 | 15 | 14 | 18 | 12 | 13 | 19 | 19 | 16 | 14 | 14 | 15 | 17 | 16 | 13 | 16 | 15 | 15 | 14 | 16 | 17 | 13 | 16 | 14 | 15 | 16 | 14 | 12 | 12 | 17
Not Completed | 3 | 4 | 1 | 4 | 2 | 1 | 3 | 2 | 3 | 1 | 1 | 2 | 3 | 4 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 0 | 4 | 3 | 2 | 0 | 3 | 2 | 5 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1, 26Wks, Counseling, CAM, AutoCalls, Feedback | 2, 26Wks, Counseling, CAM, AutoCalls, No Feedback | 3, 26Wks, Counseling, CAM, No AutoCalls, Feedback | 4, 26Wks, Counseling, CAM, No AutoCalls, No Feedback | 5, 26Wks, Counseling, No CAM, AutoCalls, Feedback | 6, 26Wks, Counseling, No CAM, AutoCalls, No Feedback | 7, 26Wks, Counseling, No CAM, No AutoCalls, Feedback | 8, 26Wks, Counseling, No CAM, No AutoCalls, No Feedback | 9, 26Wks, No Counseling, CAM, AutoCalls, Feedback | 10, 26Wks, No Counseling, CAM, AutoCalls, No Feedback | 11, 26Wks, No Counseling, CAM, No AutoCalls, Feedback | 12, 26Wks, No Counseling, CAM, No AutoCalls, No Feedback | 13, 26Wks, No Counseling, No CAM, AutoCalls, Feedback | 14, 26Wks, No Counseling, No CAM, AutoCalls, No Feedback | 15, 26Wks, No Counseling, No CAM, No AutoCalls, Feedback | 16, 26Wks, No Counseling, No CAM, No AutoCalls, No Feedback | 17, 8Wks, Counseling, CAM, AutoCalls, Feedback | 18, 8Wks, Counseling, CAM, AutoCalls, No Feedback | 19, 8Wks, Counseling, CAM, No AutoCalls, Feedback | 20, 8Wks, Counseling, CAM, No AutoCalls, No Feedback | 21, 8Wks, Counseling, No CAM, AutoCalls, Feedback | 22, 8Wks, Counseling, No CAM, AutoCalls, No Feedback | 23, 8Wks, Counseling, No CAM, No AutoCalls, Feedback | 24, 8Wks, Counseling, No CAM, No AutoCalls, No Feedback | 25, 8Wks, No Counseling, CAM, AutoCalls, Feedback | 26, 8Wks, No Counseling, CAM, AutoCalls, No Feedback | 27, 8Wks, No Counseling, CAM, No AutoCalls, Feedback | 28, 8Wks, No Counseling, CAM, No AutoCalls, No Feedback | 29, 8Wks, No Counseling, No CAM, AutoCalls, Feedback | 30, 8Wks, No Counseling, No CAM, AutoCalls, No Feedback | 31, 8Wks, No Counseling, No CAM, No AutoCalls, Feedback | 32, 8Wks, No Counseling, No CAM, No AutoCalls, No Feedback | Total
Number analyzed (Participants) | 13 | 17 | 14 | 19 | 16 | 19 | 15 | 15 | 22 | 20 | 17 | 16 | 17 | 19 | 18 | 18 | 14 | 16 | 17 | 18 | 17 | 16 | 21 | 16 | 18 | 14 | 18 | 18 | 19 | 15 | 14 | 18 | 544
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Between 18 and 65 years | 12 | 16 | 13 | 16 | 15 | 18 | 14 | 15 | 18 | 19 | 17 | 15 | 17 | 18 | 14 | 15 | 10 | 15 | 16 | 16 | 15 | 12 | 16 | 16 | 17 | 14 | 16 | 17 | 19 | 14 | 12 | 16 | 493
  >=65 years | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 4 | 3 | 3 | 1 | 1 | 2 | 2 | 4 | 5 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.08 (12.37) | 43.82 (9.87) | 39.86 (10.54) | 49.42 (14.25) | 48.81 (14.61) | 48.89 (9.72) | 47.33 (9.83) | 43.53 (8.32) | 51.55 (13.51) | 46.50 (11.04) | 44.29 (10.71) | 46.69 (11.44) | 46.41 (9.56) | 44.58 (13.68) | 49.33 (17.49) | 50.39 (12.56) | 49.07 (16.28) | 47.00 (13.11) | 42.53 (12.86) | 45.72 (12.91) | 47.35 (12.80) | 51.81 (13.97) | 48.76 (14.45) | 39.19 (11.64) | 45.50 (12.71) | 41.50 (10.71) | 42.67 (14.20) | 45.72 (10.60) | 39.53 (12.25) | 45.33 (12.69) | 47.21 (16.61) | 46.78 (13.12) | 46.12 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 8 | 12 | 11 | 13 | 9 | 9 | 12 | 11 | 9 | 11 | 11 | 10 | 10 | 10 | 8 | 9 | 10 | 10 | 11 | 10 | 12 | 10 | 11 | 8 | 10 | 10 | 12 | 9 | 8 | 11 | 321
  Male | 7 | 7 | 6 | 7 | 5 | 6 | 6 | 6 | 10 | 9 | 8 | 5 | 6 | 9 | 8 | 8 | 6 | 7 | 7 | 8 | 6 | 6 | 9 | 6 | 7 | 6 | 8 | 8 | 7 | 6 | 6 | 7 | 223
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 14 | 19 | 16 | 19 | 15 | 15 | 22 | 20 | 17 | 16 | 17 | 19 | 18 | 18 | 14 | 16 | 17 | 18 | 17 | 16 | 21 | 16 | 18 | 14 | 18 | 18 | 19 | 15 | 14 | 18 | 544

OUTCOME MEASURES:

1. Secondary Outcome: Latency to Relapse
Description: Latency to Relapse during the first 12 months post-quit, with relapse defined as 7 consecutive days of smoking; this outcome will be analyzed in a Cox regression survival analysis model with non-relapsers coded as right-censored
Time Frame: Assessed during the first 12 months post-quit after target quit day
Measure: Number; unit: participants
Groups:
- 8 Weeks of Nicotine Patch and Nicotine Gum: Participants randomized to this condition received 8 Weeks of Nicotine Patch and Nicotine Gum; participants in this group received all combinations of the other four study treatments: No Maintenance Counseling or Maintenance Counseling; No Cognitive Medication Adherence Counseling (C-MAC) or C-MAC; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The 8 Weeks of Nicotine Patch and Nicotine Gum group consists of 269 participants (approximately half the total sample of 544) who will be compared with a group that received 26 Weeks of Nicotine Patch and Nicotine Gum (N=275; approximately half the total sample) in a main effect statistical comparison (8 Weeks of Nicotine Patch and Nicotine Gum vs. 26 Weeks of Nicotine Patch and Nicotine Gum).
- 26 Weeks of Nicotine Patch and Nicotine Gum: Participants randomized to this condition received 26 Weeks of Nicotine Patch and Nicotine Gum; participants in this group received all combinations of the other four study treatments: No Maintenance Counseling or Maintenance Counseling; No Cognitive Medication Adherence Counseling (C-MAC) or C-MAC; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The 26 Weeks of Nicotine Patch and Nicotine Gum group consists of 275 participants (approximately half the total sample of 544) who will be compared with a group that received 8 Weeks of Nicotine Patch and Nicotine Gum (N=269; approximately half the total sample) in a main effect statistical comparison (8 Weeks of Nicotine Patch and Nicotine Gum vs. 26 Weeks of Nicotine Patch and Nicotine Gum).
- No Maintenance Counseling: Participants randomized to this condition received No Maintenance Counseling; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Cognitive Medication Adherence Counseling (C-MAC) or C-MAC; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The No Maintenance Counseling group consists of 281 participants (approximately half the total sample of 544) who will be compared with a group that received Maintenance Counseling (N=263; approximately half the total sample) in a main effect statistical comparison (No Maintenance Counseling vs. Maintenance Counseling).
- Maintenance Counseling: Participants randomized to this condition received Maintenance Counseling; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Cognitive Medication Adherence Counseling (C-MAC) or C-MAC; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The Maintenance Counseling group consists of 263 participants (approximately half the total sample of 544) who will be compared with a group that received Maintenance Counseling (N=281; approximately half the total sample) in a main effect statistical comparison (No Maintenance Counseling vs. Maintenance Counseling).
- No Cognitive Medication Adherence Counseling: Participants randomized to this condition received No Cognitive Medication Adherence Counseling; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Maintenance Counseling or Maintenance Counseling; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The No Cognitive Medication Adherence Counseling group consists of 273 participants (approximately half the total sample of 544) who will be compared with a group that received Cognitive Medication Adherence Counseling (N=271; approximately half the total sample) in a main effect statistical comparison (No Cognitive Medication Adherence Counseling vs. Cognitive Medication Adherence Counseling).
- Cognitive Medication Adherence Counseling: Participants randomized to this condition received Cognitive Medication Adherence Counseling; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Maintenance Counseling or Maintenance Counseling; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The Cognitive Medication Adherence Counseling group consists of 271 participants (approximately half the total sample of 544) who will be compared with a group that received No Cognitive Medication Adherence Counseling (N=273; approximately half the total sample) in a main effect statistical comparison (No Cognitive Medication Adherence Counseling vs. Cognitive Medication Adherence Counseling).
- Electronic Medication Monitoring Device Without Feedback: Participants randomized to this condition received an Electronic Medication Monitoring Device Without Feedback; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Maintenance Counseling or Maintenance Counseling; No Cognitive Medication Adherence Counseling or Cognitive Medication Adherence Counseling; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The Electronic Medication Monitoring Device Without Feedback group consists of 274 participants (approximately half the total sample of 544) who will be compared with a group that received an Electronic Medication Monitoring Device Plus Feedback (N=270; approximately half the total sample) in a main effect statistical comparison (Electronic Medication Monitoring Device Without Feedback vs. Electronic Medication Monitoring Device Plus Feedback).
- Electronic Medication Monitoring Device Plus Feedback: Participants randomized to this condition received an Electronic Medication Monitoring Device Plus Feedback; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Maintenance Counseling or Maintenance Counseling; No Cognitive Medication Adherence Counseling or Cognitive Medication Adherence Counseling; No Automated Adherence Prompting Phone Calls or Automated Adherence Prompting Phone Calls. The Electronic Medication Monitoring Device Plus Feedback group consists of 270 participants (approximately half the total sample of 544) who will be compared with a group that received an Electronic Medication Monitoring Device Without Feedback (N=274; approximately half the total sample) in a main effect statistical comparison (Electronic Medication Monitoring Device Without Feedback vs. Electronic Medication Monitoring Device Plus Feedback).
- No Automated Adherence Prompting Phone Calls: Participants randomized to this condition received No Automated Adherence Prompting Phone Calls; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Maintenance Counseling or Maintenance Counseling; No Cognitive Medication Adherence Counseling or Cognitive Medication Adherence Counseling; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback. The No Automated Adherence Prompting Phone Calls group consists of 272 participants (approximately half the total sample of 544) who will be compared with a group that received Automated Adherence Prompting Phone Calls (N=272; approximately half the total sample) in a main effect statistical comparison (No Automated Adherence Prompting Phone Calls vs. Automated Adherence Prompting Phone Calls).
- Automated Adherence Prompting Phone Calls: Participants randomized to this condition received Automated Adherence Prompting Phone Calls; participants in this group received all combinations of the other four study treatments: 8 Weeks of Nicotine Patch and Nicotine Gum or 26 Weeks of Nicotine Patch and Nicotine Gum; No Maintenance Counseling or Maintenance Counseling; No Cognitive Medication Adherence Counseling or Cognitive Medication Adherence Counseling; Electronic Medication Monitoring Device Without Feedback or Electronic Medication Monitoring Device Plus Feedback. The Automated Adherence Prompting Phone Calls group consists of 272 participants (approximately half the total sample of 544) who will be compared with a group that received No Automated Adherence Prompting Phone Calls (N=272; approximately half the total sample) in a main effect statistical comparison (No Automated Adherence Prompting Phone Calls vs. Automated Adherence Prompting Phone Calls).
Arm/Group | 8 Weeks of Nicotine Patch and Nicotine Gum | 26 Weeks of Nicotine Patch and Nicotine Gum | No Maintenance Counseling | Maintenance Counseling | No Cognitive Medication Adherence Counseling | Cognitive Medication Adherence Counseling | Electronic Medication Monitoring Device Without Feedback | Electronic Medication Monitoring Device Plus Feedback | No Automated Adherence Prompting Phone Calls | Automated Adherence Prompting Phone Calls
Number analyzed (Participants) | 269 | 275 | 281 | 263 | 273 | 271 | 274 | 270 | 272 | 272
participants
  # Participants Who Relapsed (Smoking) | 227 | 209 | 228 | 208 | 214 | 222 | 225 | 211 | 218 | 218
  # Participants Who Did Not Relapse (Not Smoking) | 42 | 66 | 53 | 55 | 59 | 49 | 49 | 59 | 54 | 54
Statistical Analysis 1: Comparison: 8 Weeks of Nicotine Patch and Nicotine Gum vs 26 Weeks of Nicotine Patch and Nicotine Gum; The Cox regression model effects consisted of five treatment effects, 10 two-way treatment interactions, 10 three-way treatment interactions, and two covariates : two items from the Fagerstrom Test of Nicotine Dependence (Item 1: time to first cigarette; Item 4: cigarettes per day); Test type: Superiority or Other; p = .045, Regression, Cox; Cox Proportional Hazard = .906, 95% CI 2-sided [.822 to .998]
Statistical Analysis 2: Comparison: No Maintenance Counseling vs Maintenance Counseling; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .705, Regression, Cox; Cox Proportional Hazard = .982, 95% CI 2-sided [.892 to 1.081]
Statistical Analysis 3: Comparison: No Cognitive Medication Adherence Counseling vs Cognitive Medication Adherence Counseling; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .382, Regression, Cox; Cox Proportional Hazard = 1.044, 95% CI 2-sided [.948 to 1.149]
Statistical Analysis 4: Comparison: Electronic Medication Monitoring Device Without Feedback vs Electronic Medication Monitoring Device Plus Feedback; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .339, Regression, Cox; Cox Proportional Hazard = .954, 95% CI 2-sided [.867 to 1.050]
Statistical Analysis 5: Comparison: No Automated Adherence Prompting Phone Calls vs Automated Adherence Prompting Phone Calls; Test type: Superiority or Other; p = .248, Regression, Cox; Cox Proportional Hazard = .945, 95% CI 2-sided [.858 to 1.040]

2. Primary Outcome: Self-Reported 7-Day Point-Prevalence Abstinence
Description: Self-Reported 7-Day Point-Prevalence Abstinence is a dichotomous outcome with values of 0 and 1 where 0=smoking on one or more of the past 7 days at the assessment endpoint (52 weeks post-quit) and 1=no smoking on any of the past 7 days at the assessment endpoint (i.e., abstinent for the past 7 days); this outcome will be analyzed in a logistic regression analysis model.
  Note: This abstinence primary outcome replaces latency to relapse (now designated as a secondary outcome) because reviewers of the now-accepted manuscript (at the journal "Addiction") advised us to change the primary outcome to the current week 52 Self-Reported 7-Day Point-Prevalence Abstinence.
Time Frame: Assessed at 52 weeks after target quit day
Measure: Number; unit: participants
Arm/Group | 8 Weeks of Nicotine Patch and Nicotine Gum | 26 Weeks of Nicotine Patch and Nicotine Gum | No Maintenance Counseling | Maintenance Counseling | No Cognitive Medication Adherence Counseling | Cognitive Medication Adherence Counseling | Electronic Medication Monitoring Device Without Feedback | Electronic Medication Monitoring Device Plus Feedback | No Automated Adherence Prompting Phone Calls | Automated Adherence Prompting Phone Calls
Number analyzed (Participants) | 269 | 275 | 281 | 263 | 273 | 271 | 272 | 272 | 274 | 270
participants
  # Participants Who Smoking | 197 | 181 | 202 | 176 | 184 | 194 | 186 | 192 | 198 | 180
  # Participants Who Are Abstinent | 72 | 94 | 79 | 87 | 89 | 77 | 86 | 80 | 76 | 90
Statistical Analysis 1: Comparison: 8 Weeks of Nicotine Patch and Nicotine Gum vs 26 Weeks of Nicotine Patch and Nicotine Gum; The logistic regression model effects consisted of five treatment main effects and all treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., 8 Weeks of Nicotine Patch and Nicotine Gum vs. 26 Weeks of Nicotine Patch and Nicotine Gum) would result in significantly higher abstinence at 52 weeks after target quit day; Test type: Superiority or Other; p = .011, Regression, Logistic; Odds Ratio (OR) = 1.402, 95% CI 2-sided [1.080 to 1.821]
Statistical Analysis 2: Comparison: No Maintenance Counseling vs Maintenance Counseling; The logistic regression model effects consisted of five treatment main effects and all treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., No Maintenance Counseling vs. Maintenance Counseling) would result in significantly higher abstinence at 52 weeks after target quit day; Test type: Superiority or Other; p = .956, Regression, Logistic; Odds Ratio (OR) = 1.008, 95% CI 2-sided [.769 to 1.321]
Statistical Analysis 3: Comparison: No Cognitive Medication Adherence Counseling vs Cognitive Medication Adherence Counseling; The logistic regression model effects consisted of five treatment main effects and all treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., No Cognitive Medication Adherence Counseling vs. Cognitive Medication Adherence Counseling) would result in significantly higher abstinence at 52 weeks after target quit day; Test type: Superiority or Other; p = .885, Regression, Logistic; Odds Ratio (OR) = 1.018, 95% CI 2-sided [.797 to 1.301]
Statistical Analysis 4: Comparison: Electronic Medication Monitoring Device Without Feedback vs Electronic Medication Monitoring Device Plus Feedback; The logistic regression model effects consisted of five treatment main effects and all treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., Electronic Medication Monitoring Device Without Feedback vs. Electronic Medication Monitoring Device Plus Feedback) would result in significantly higher abstinence at 52 weeks after target quit day; Test type: Superiority or Other; p = .205, Regression, Logistic; Odds Ratio (OR) = .852, 95% CI 2-sided [.664 to 1.092]
Statistical Analysis 5: Comparison: No Automated Adherence Prompting Phone Calls vs Automated Adherence Prompting Phone Calls; The logistic regression model effects consisted of five treatment main effects and all treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., No Automated Adherence Prompting Phone Calls vs. Automated Adherence Prompting Phone Calls) would result in significantly higher abstinence at 52 weeks after target quit day; Test type: Superiority or Other; p = .514, Regression, Logistic; Odds Ratio (OR) = 1.090, 95% CI 2-sided [.842 to 1.411]

ADVERSE EVENTS:
Time Frame: AEs were reported for 8 or 26 weeks (for the duration of time when the participant was on medication.)
Description: Protocol prompted AE assessments occurred at weeks 1, 4, 8 (and 16 for those on medication for 16 weeks) postquit. Data from ad Hoc AE reports and protocol prompted AE assessments were combined. Only AEs where 5% or more of those from a study arm were reported and compared to other study arms.
Groups:
- 26 Weeks of Nicotine Patch and Nicotine Gum: Participants randomized to this condition received 26 Weeks of Nicotine Patch and Nicotine Gum.
  IF the participant smoked >10 cigs/day AND is randomized to a 26 week medication condition: they were asked to take one 21 mg patch per day for 22 weeks, THEN one 14 mg patch per day for 2 weeks, THEN one patch 7 mg patch per day for 2 weeks. Participants were also asked to use one piece of one 4-mg- gum every 1-2 hours (9 pieces maximum per day)for 24 weeks and decrease gum use over the 2 weeks prior to medication termination until they are down to one gum piece every 4-8 hours by the last week of treatment.
  IF the participant smoked 5-10 cigs/day AND is randomized to a 26 week medication condition: they were asked to take one 14 mg patch per day for 22 weeks, THEN one patch 7 mg patch per day for 4 weeks. Participants were also asked to use one piece of 2-mg gum every 1-2 hours (9 pieces maximum per day)for 24 weeks and decrease gum use over the 2 weeks prior to medication
- 8 Weeks of Nicotine Patch and Nicotine Gum: Participants randomized to this condition received 8 Weeks of Nicotine Patch and Nicotine Gum.
  IF participant smoked >10 cigs/day AND is randomized to a 8 week condition: they were asked to take one 21 mg patch/day for 4 weeks, THEN one 14 mg patch/day for 2 weeks, THEN one patch 7mg/day for 2 weeks.Participants were also asked to use 4-mg gum every 1-2 hours (9 pieces maximum per day)for 6 weeks and decrease gum use over the 2 weeks prior to medication termination until down to one gum piece every 4-8 hours by the last week of treatment.
  IF participant smoked 5-10 cigs/day AND is randomized to the 8 week medication condition: they were asked to take one 14 mg patch/day for 4 weeks, THEN one 7 mg patch/day for 4 weeks. Participants were also asked to use 2-mg gum every 1-2 hours (9 pieces max per day)for 6 weeks and decrease gum use over the 2 weeks prior to medication termination until down to one gum piece every 4-8 hours by the last week of treatment.
Arm/Group | 26 Weeks of Nicotine Patch and Nicotine Gum | 8 Weeks of Nicotine Patch and Nicotine Gum
Serious Adverse Events (participants affected / at risk) | 10/275 | 6/269
Other Adverse Events (participants affected / at risk) | 146/275 | 141/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 26 Weeks of Nicotine Patch and Nicotine Gum (N=275) | 8 Weeks of Nicotine Patch and Nicotine Gum (N=269)
Cardiovascular (Cardiac disorders) | 4 (4) | 5 (6)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death-unknown cause (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 26 Weeks of Nicotine Patch and Nicotine Gum (N=275) | 8 Weeks of Nicotine Patch and Nicotine Gum (N=269)
Dizziness (Nervous system disorders) | 23 | 19
Headache (Nervous system disorders) | 24 | 19
Indigestion (Gastrointestinal disorders) | 28 | 28
Insomnia (Nervous system disorders) | 29 | 31
Itches or Hives (Skin and subcutaneous tissue disorders) | 28 | 18
Mouth Problems (Gastrointestinal disorders) | 17 | 18
Nausea (Gastrointestinal disorders) | 40 | 39
Skin Rash (Skin and subcutaneous tissue disorders) | 63 | 50
VividDreams (Nervous system disorders) | 44 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes